CLINICAL TRIAL: NCT06205511
Title: The Prevalence of Oral HPV Infection and Oral Lesions in People Living With HIV in a HIV Primary Care Clinic
Brief Title: The Prevalence of Oral HPV Infection and Oral Lesions in People Living With HIV
Acronym: SWISH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vivent Health (Other)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Principal Investigator, Cindy Firnhaber, MD, Director of Research, Vivent Health
Other Study IDs: MISP #10965
Record Dates: First submitted 2023-05-03; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-09

CONDITIONS: Human Immunodeficiency Virus; Human Papilloma Virus
Keywords: HPV; HIV; SWISH
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Group: Single group, observational cross-sectional cohort.
  Interventions: Diagnostic Test: Oral HPV Sample

INTERVENTIONS:
Diagnostic Test: Oral HPV Sample — The study participant will be asked to provide an oral swish and spit sample. This sample collection will follow the procedure published by (Herrero et al 2013). The specimen is collected by a 15-second rinse followed by a 15-second gargle using 15 ml of an alcohol-based mouth wash such as a commercially available product, Scope. The 15-ml samples will then be stored at -20 and then shipped on dry ice to Dr. Anna Giuliano's laboratory in Tampa Florida for HPV testing. At present Dr. Giuliano's laboratory is using the DDL SPF10 LiPA assay for sample analysis. An oral exam will be performed for each patient by the Vivent Dentist within 30 days of the collection of the HPV sample. If a referral is needed to an oral surgeon or Ears, Nose, and Throat specialist this will be done within 60 days of the dentist visit. The HPV results will not be shared with the participants as these are research study results and not part of standard of care.

SUMMARY:
The study will evaluate 300 people living with HIV that attend the Vivent Clinic for HIV care. We will characterize our population and include age, race/ethnicity, sex at birth, tobacco use, alcohol use, other comorbidities, HPV vaccination status, other HPV disease, and lab values such as CD4 count and HIV viral load. We will compare results between participants who are HPV positive and negative. We will also evaluate the relationship between HPV oral infections and lesions and the variables above to better understand possible predictors of HPV infections and lesions.

DETAILED DESCRIPTION:
Vivent Health is a non-profit medical home model dedicated to the primary care of People Living with HIV (PLWH) and also provides pre-exposure prophylaxis (PrEP), Hepatitis C, and sexually transmitted infection (STI) treatment. The organization has clinics in Wisconsin (multiple cities), Denver, St. Louis, Austin and Kansas City. All insurances except Kaiser are honored and non-insured people are able to be seen. The Denver medical clinic is a designated medical home that provides adult primary medical and specialty care to approximately 1000 + PLWH. In additional to medical care, this clinic has an onsite pharmacy, case management, HIV and Hepatitis C prevention department, syringe access program, legal department, housing specialists, food bank, a mental health program and dental services. Vivent Health in Denver cares for a diverse population with approximately 11% African-American, 13% Latino, and a recently increasing percentage of women around 13%. This clinic has a strong Electronic Health Record System (EHR- Epic) which provides ample opportunity to recruit a robust study population to investigate the following co-morbidities which might increase the risk of oral HPV infection and related lesions. Given the lack of recommended routine screening for oral HPV in the absence of established masses or lesions, there is a wealth of opportunities to investigate risk factors associated with the presence and prevalence of oral HPV which, in turn, can potentially be used to inform screening and treatment protocols. This proposal is designed to evaluate the prevalence of oral HPV infections and associated oral lesions and associated demographics in HIV treatment clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV test on any FDA-approved HIV test
2. Ability and willingness of participant to provide informed consent
3. Capable of performing an oral swish and spit sample collection
4. Willingness to have an oral exam by Denver Vivent Health Dentist
5. Has had at least two visits at the Vivent Health Denver clinic
6. Study participant allows demographics and medical history/laboratory results in electronic medical records to be confidentially evaluated.

Exclusion Criteria:

1. Any medical or mental health diagnosis that the study team concludes would prohibits participation of the protocol
2. CD4 count < 200 cells/ml
3. History of Oral/tongue cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive patients of the Vivent Health Denver clinic.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
HPV Prevalence in people living with HIV | single visit study for participants and will collect 300 oral samples at the visit and will analyze samples and statistics after completion of enrolling 300 participants in approximately 18 months from the start study
  To evaluate the prevalence of positive oral HPV in a population of PLWH and to compare prevalence rate with the historically documented prevalence rates in the general population

SECONDARY OUTCOMES:
Demographics of other factors to oral HPV | This is a single visit study for participants and will collect 300 oral samples at the visit and will analyze samples and will compare participant demographics with HIV disease state in approximately 18 months from the start study
  To evaluate the correlation of HIV disease factors and demographics in study participatants including CD4 nadir, recent CD4, recent viral load, sexual activity, HPV vaccination status , age, sex, and race compared to participants with samples that are positive for oral HPV
Correlation of other factors to oral HPV | This is a single visit study for participants analyze samples and participant demographic in approximately 18 months from the start study
  To evaluate the correlation of factors including CD4 nadir, recent CD4, recent viral load, sexual activity, HPV vaccination status, age, sex, and race with the prevalence of oral HPV
Oral lesion prevalence with HPV positive samples | This is a single visit study for participants and will analyze samples and participant demographics with any oral lesions in approximately 18 months from the start study
  To evaluate the prevalence of oral lesions in patients who test positive for oral HPV through screening

CONTACTS AND LOCATIONS:
Locations (1):
- Vivent Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time no plan to share IPD has been created, but might be a path considered in the future if requested

REFERENCES:
- [Background] Chaturvedi AK, Graubard BI, Broutian T, Pickard RKL, Tong ZY, Xiao W, Kahle L, Gillison ML. Effect of Prophylactic Human Papillomavirus (HPV) Vaccination on Oral HPV Infections Among Young Adults in the United States. J Clin Oncol. 2018 Jan 20;36(3):262-267. doi: 10.1200/JCO.2017.75.0141. Epub 2017 Nov 28. PMID 29182497
- [Background] Deeken JF, Tjen-A-Looi A, Rudek MA, Okuliar C, Young M, Little RF, Dezube BJ. The rising challenge of non-AIDS-defining cancers in HIV-infected patients. Clin Infect Dis. 2012 Nov;55(9):1228-35. doi: 10.1093/cid/cis613. Epub 2012 Jul 9. PMID 22776851
- [Background] Grulich AE, van Leeuwen MT, Falster MO, Vajdic CM. Incidence of cancers in people with HIV/AIDS compared with immunosuppressed transplant recipients: a meta-analysis. Lancet. 2007 Jul 7;370(9581):59-67. doi: 10.1016/S0140-6736(07)61050-2. PMID 17617273
- [Background] Patel P, Hanson DL, Sullivan PS, Novak RM, Moorman AC, Tong TC, Holmberg SD, Brooks JT; Adult and Adolescent Spectrum of Disease Project and HIV Outpatient Study Investigators. Incidence of types of cancer among HIV-infected persons compared with the general population in the United States, 1992-2003. Ann Intern Med. 2008 May 20;148(10):728-36. doi: 10.7326/0003-4819-148-10-200805200-00005. PMID 18490686
- [Background] McQuillan G, Kruszon-Moran D, Markowitz LE, Unger ER, Paulose-Ram R. Prevalence of HPV in Adults Aged 18-69: United States, 2011-2014. NCHS Data Brief. 2017 Apr;(280):1-8. PMID 28463105
- [Background] Rodriguez AC, Schiffman M, Herrero R, Wacholder S, Hildesheim A, Castle PE, Solomon D, Burk R; Proyecto Epidemiologico Guanacaste Group. Rapid clearance of human papillomavirus and implications for clinical focus on persistent infections. J Natl Cancer Inst. 2008 Apr 2;100(7):513-7. doi: 10.1093/jnci/djn044. Epub 2008 Mar 25. PMID 18364507
- [Background] Plummer M, Schiffman M, Castle PE, Maucort-Boulch D, Wheeler CM; ALTS Group. A 2-year prospective study of human papillomavirus persistence among women with a cytological diagnosis of atypical squamous cells of undetermined significance or low-grade squamous intraepithelial lesion. J Infect Dis. 2007 Jun 1;195(11):1582-9. doi: 10.1086/516784. Epub 2007 Apr 16. PMID 17471427
- [Background] Shiels MS, Althoff KN, Pfeiffer RM, Achenbach CJ, Abraham AG, Castilho J, Cescon A, D'Souza G, Dubrow R, Eron JJ, Gebo K, John Gill M, Goedert JJ, Grover S, Hessol NA, Justice A, Kitahata M, Mayor A, Moore RD, Napravnik S, Novak RM, Thorne JE, Silverberg MJ, Engels EA; North American AIDS Cohort Collaboration on Research and Design (NA-ACCORD) of the International Epidemiologic Databases to Evaluate AIDS (IeDEA). HIV Infection, Immunosuppression, and Age at Diagnosis of Non-AIDS-Defining Cancers. Clin Infect Dis. 2017 Feb 15;64(4):468-475. doi: 10.1093/cid/ciw764. PMID 27940936
- [Background] Van Dyne EA, Henley SJ, Saraiya M, Thomas CC, Markowitz LE, Benard VB. Trends in Human Papillomavirus-Associated Cancers - United States, 1999-2015. MMWR Morb Mortal Wkly Rep. 2018 Aug 24;67(33):918-924. doi: 10.15585/mmwr.mm6733a2. PMID 30138307
- [Background] Vokes EE, Agrawal N, Seiwert TY. HPV-Associated Head and Neck Cancer. J Natl Cancer Inst. 2015 Dec 9;107(12):djv344. doi: 10.1093/jnci/djv344. Print 2015 Dec. PMID 26656751
- [Background] Herrero R, Quint W, Hildesheim A, Gonzalez P, Struijk L, Katki HA, Porras C, Schiffman M, Rodriguez AC, Solomon D, Jimenez S, Schiller JT, Lowy DR, van Doorn LJ, Wacholder S, Kreimer AR; CVT Vaccine Group. Reduced prevalence of oral human papillomavirus (HPV) 4 years after bivalent HPV vaccination in a randomized clinical trial in Costa Rica. PLoS One. 2013 Jul 17;8(7):e68329. doi: 10.1371/journal.pone.0068329. Print 2013. PMID 23873171

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT06205511/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT06205511/ICF_001.pdf